CLINICAL TRIAL: NCT04327440
Title: Combined Effects of RTS,S Vaccination and PBO Nets on Malaria Infection and Transmission in Malawi
Brief Title: RTSS Vaccine and PBO Net Impact on Malaria Infection and Transmission in Malawi
Acronym: RTSS/PBO
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); University of Maryland, Baltimore (Other); Boston University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Terrie Taylor, Professor, Michigan State University
Other Study IDs: 00002662; 3U19AI089683-10S1 (NIH)
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Malaria, Malaria Vaccine, Insecticide-treated Bednets
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots to identify malaria infection (asexual parasites) and transmission potential (sexual stage parasites).
  Plasma to assess serological measures of exposure and antimalarial immunity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nyambi, rainy season: 250 children of age-eligible for RTS,S vaccine (7-18 months) 500 siblings (>18 months, < 10 years of age)
  The duration of the cohort is six months.
  Interventions: Biological: RTS,S/AS01 malaria vaccine; Other: PBO bed nets
- Nyambi, dry season: 250 children of age-eligible for RTS,S vaccine (7-18 months) 500 siblings (>18 months, < 10 years of age)
  The duration of the cohort is six months.
  Interventions: Biological: RTS,S/AS01 malaria vaccine; Other: PBO bed nets
- Kalembo, rainy season: 250 children of age-eligible for RTS,S vaccine (7-18 months) 500 siblings (>18 months, < 10 years of age)
  The duration of the cohort is six months.
- Kalembo, dry season: 250 children of age-eligible for RTS,S vaccine (7-18 months) 500 siblings (>18 months, < 10 years of age)
  The duration of the cohort is six months.

INTERVENTIONS:
Biological: RTS,S/AS01 malaria vaccine — Malaria vaccine: RTS,S is a subunit vaccine that includes a portion of the circumsporozoite protein (CSP) co-expressed with Hepatitis B surface antigen combined with an adjuvant. The Phase 3 trial of three doses administered to 5-17-month-olds confirmed moderate protection, with overall efficacy estimates of 50.4% against clinical malaria and 34.8% against severe malaria after three doses. Efficacy, which waned over time, was marginally improved by boosting at 18 months. The European Medicines Agency adopted a positive scientific opinion of the vaccine for use outside of the European Union. The World Health Organization has created the Malaria Vaccine Implementation Program (MVIP) and selected Malawi as one of the sites to explore the feasibility, efficacy and safety of RTS,S vaccination in the context of routine use.
  Other Names: RTS,S
  Groups: Nyambi, dry season; Nyambi, rainy season
Other: PBO bed nets — PBO nets: The PBO nets represent a new formulation of insecticide-treated bed nets with a chemical synergist, piperonyl butoxide (PBO), designed to enhance the insecticidal effect of pyrethroids. They seem to be helpful in areas like Malawi where insecticide-resistance is increasing. PBO inhibits the enzyme that detoxifies the pyrethroid, allowing the pyrethroid to act on the mosquito. The impact of PBO net use was also detectable in key entomological measures including Anopheles density, sporozoite rate and entomological inoculation rates. Following these promising preliminary results in Tanzania, Malawi's National Malaria Control Program (NMCP) is piloting the use of PBO-nets iin one of our two study sites, presenting us with the opportunity to study the effectiveness of these nets in the context of real-world program setting
  Groups: Nyambi, dry season; Nyambi, rainy season

SUMMARY:
The overall goal of this study is to assess the impact of RTS,S (malaria) vaccination and PBO nets on malaria infection and transmission, independently and how they interact when they are introduced together.

The specific objectives for the study are as follows:

1. To estimate the impact of PBO nets and RTS,S vaccine on Plasmodium infection prevalence and transmission, independently and how they interact when they are introduced together in Malawi (Phase 1).
2. To assess the feasibility of evaluating the impact of RTS,S vaccine and PBO nets independently in a larger scale future study.

DETAILED DESCRIPTION:
Introduction: The decline in malaria incidence has stalled globally and incidence is increasing in some high transmission settings of sub-Saharan Africa, including Malawi. The situation is worsening despite the scale-up of previously effective interventions, raising concerns that the impact of current malaria control and prevention strategies maybe compromised.

Problem: There is an urgent need for innovative approaches to malaria control and Malawi is currently positioned to assess two of the most promising new interventions. The Malawi Ministry of Health (MOH) is launching large scale projects to evaluate a new formulation of insecticide-treated bed nets with a chemical synergist, piperonyl butoxide (PBO), designed to enhance the insecticidal effect of pyrethroids and the new malaria vaccine RTS,S (RTS,S). In an effort to gain the most information from these, interventions Malawi's National Malaria Control Programme (NMCP) have invited the Malawi International Center for Excellence in Malaria Research (ICEMR) to evaluate the effectiveness of the two interventions (alone and in combination) on malaria prevalence and transmission.

Objective: In this proposed implementation study, we propose to assess the impact of PBO nets and RTS,S vaccine on Plasmodium infection prevalence and transmission.

Study type and methodology: We will enroll children in a prospective cohort study in which the follow-up will be at the 2nd, 4th, and 6th month. We are selecting two health center catchment areas: one in which both RTS,S and PBO nets are available through the government health system and one in which there is no RTS,S vaccine available and standard long-lasting insecticide-treated nets (LLINS) have been distributed through the public section. At each visit, we will collect specimens to identify malaria infection and detect gametocyte infections. We will also collect and analyze mosquitoes from 100 households in both catchment areas to provide an entomological evidence of the force of infection. Children in households that are scheduled to receive both PBO nets and RTS,S vaccine will be compared to children in households that are not scheduled to receive either of these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 18 months of age (age-eligible for at least 3 doses of RTS,S doses) OR being one of not more than two children living in the household of an enrolled age-eligible child and being >18 mos and < 10 years of age.
* Not on cotrimoxazole prophylaxis for HIV infection
* Weight >5 kg
* Permanent residence of Health Centre (HC) catchment area
* Residence within 10 km from the HC
* Written informed consent from parent/guardian for the child to participate in the study

Exclusion Criteria:

Non-residents of the catchment area and visitors to the study area will be excluded because the study requires follow-up for at least 6 months and access to interventions such as conventional, PBO nets and malaria vaccination.

Ages: 7 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children whose age is between 7 and 18 months, which indicates they could receive at least 3 RTS,S doses, will be eligible to participate. Following informed consent from parents/guardians, up to two children who are 18 months but ≤10 years of age, from the same household as the vaccine-eligible child, will also be enrolled. Only households whose families intend to stay in the area for at least six months and whose eligible children will also be expected to use an assigned health center for child vaccinations will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 1691 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Malaria infection prevalence | 6 months/cohort, 4 cohorts in Phase 1
  Comparison of malaria infection prevalence in RTS/S cohorts compared to cohorts not exposed to RTS,S
Anopheles species abundance | 6 months/cohort, 4 cohorts in Phase 1
  Comparison of Anopheles captured in households with PBO nets compared to household with conventional nets

SECONDARY OUTCOMES:
Gametocyte prevalence | 6 months/cohort, 4 cohorts
  Comparison of the prevalence of gametocytes (male and female) in cohorts exposed to RTS,S vs those not exposed
Net usage | 6 months/cohort, 4 cohorts
  Comparison of nightly net usage in cohorts with PBO nets compared to cohorts with conventional nets
Serological markers of immunity and exposure | 6 months/cohort, 4 cohorts
  Comparison of serological markers in cohorts exposed to RTS,S vs those not exposed to RTS,S
Anopheles gravidity rates | 6 months/cohort, 4 cohorts
  Comparison of Anopheles gravidity rates in cohorts with PBO nets compared to cohorts with conventional nets
Anopheles sporozoite rates | 6 months/cohort, 4 cohorts
  Comparison of Anopheles sporozoite rates in cohorts with PBO nets compared to cohorts with conventional nets

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malawi College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04327440/Prot_SAP_000.pdf